CLINICAL TRIAL: NCT04964986
Title: A Multicenter, Open-label, Metabolic Balance Study to Evaluate the Effects of Apraglutide on Intestinal Absorption in Adult Subjects With Short Bowel Syndrome, Intestinal Failure (SBS-IF), and Colon-in-Continuity (CIC)
Brief Title: Metabolic Balance Study of Apraglutide in Patients With Short Bowel Syndrome, Intestinal Failure (SBS-IF) and Colon-in-Continuity (CIC)
Acronym: STARSnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA799-013; 2020-005129-99 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-07-16 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Short Bowel Syndrome
Keywords: Intestinal Failure; SBS; SBS-IF; CIC; Colon-in-Continuity
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — apraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apraglutide (Experimental): All participants received apraglutide administered subcutaneously (SC) once weekly for 52 weeks.
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Apraglutide is a synthetic peptide analogue of GLP-2 under development for treatment of SBS-IF, which acts as a full agonist at the GLP-2 receptor with in vitro potency and selectivity comparable with native GLP-2.
  Other Names: TA799

SUMMARY:
The primary objective of the trial is to evaluate the safety of apraglutide in adult subjects with SBS-IF and CIC.

DETAILED DESCRIPTION:
This is an international, multicenter trial to evaluate the safety of apraglutide in adult participants with SBS-IF and CIC. The active pharmaceutical ingredient is apraglutide, an investigational glucagon-like peptide-2 (GLP-2) analogue. The trial consists of an evaluation period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for this trial prior to any trial specific assessment.
* Male and female subjects with SBS-IF and CIC, receiving parenteral support (PS), secondary to surgical resection of the small intestine with < 200 cm from duodenojejunal flexure.
* Subject must require parenteral support (PS) at least 2 days per week and be considered stable.
* No restorative surgery intended to change PS requirements in the trial period.
* Age ≥ 18 years at screening.

Exclusion Criteria:

* Pregnancy or lactation.
* Body mass index equal or higher than 30 kg/m^2 at the time of screening.
* Major abdominal surgery in the last 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (2):
- UZ Leuven, Leuven, Belgium
- Beaujon Hospital, Clichy, France

REFERENCES:
- [Derived] Verbiest A, Hvistendahl MK, Bolognani F, Li C, Youssef NN, Huh S, Menys A, Bhatnagar G, Vanslembrouck R, Peeters R, Sartoris R, Vermeersch P, Wauters L, Verbeke K, Jeppesen PB, Joly F, Vanuytsel T. Efficacy and safety of apraglutide in short bowel syndrome with intestinal failure and colon-in-continuity: A multicenter, open-label, metabolic balance study. Clin Nutr. 2024 Dec;43(12):158-166. doi: 10.1016/j.clnu.2024.10.011. Epub 2024 Oct 16. PMID 39461299

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 10 participants with SBS-IF and CIC enrolled, 9 participants were treated and analyzed. The participant who enrolled but was not treated was not included in any study analysis.
Groups:
- Apraglutide SC Injections, Once Weekly: All participants received apraglutide administered subcutaneously (SC) once weekly for 52 weeks.
Period: Overall Study
Arm/Group | Apraglutide SC Injections, Once Weekly
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled and treated participants.
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (17.46)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 8
  65-84 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-Emergent Adverse Event (TEAE)
Description: A TEAE was any unfavorable and unintended sign, symptom, or disease temporally associated with apraglutide, whether or not related, that occurred or worsened after the dose of apraglutide. A serious TEAE was defined as any TEAE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. Clinically significant changes from baseline in clinical chemistry, hematology, hemostasis, anti-drug antibodies (ADAs), and urine analysis were reported as adverse events.
  Adverse events of special interest (AESI) included injection site reaction, gastrointestinal obstruction, gallbladder, biliary, and pancreatic disease, fluid overload, colorectal polyps, malignancies.
Time Frame: Day 1 up to approximately 55 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  At least one TEAE | 9
  At least one treatment-related TEAE | 5
  At least one TESAE | 3
  At least one treatment-related TESAE | 1
  At least one treatment-emergent AESI | 3
  At least one TEAE leading to dose interruption | 1
  At least one TEAE leading to permanent dose discontinuation | 0

2. Primary Outcome: Absolute Change in Absorption of Energy Over Metabolic Balance (MB) Periods From Baseline at Week 48
Description: Applicable to Protocol V3.0 implemented in France (classed as secondary endpoint in Protocol V4.0 [implemented in Belgium]).
  The absorption was defined as dietary intake minus output from fecal excretion over a 72-hour MB period at a given analysis time point. Since dietary intake and fecal excretion were measured daily, i.e., up to three measurements may contribute to absorption calculations, the average over all available daily absorption measurements over the 72-hour period were used for analysis.
Time Frame: Baseline and Week 48
Population: The full analysis set included all participants who received at least one dose of trial treatment and contributed at least one valid post-baseline efficacy point.
Measure: Mean (Standard Deviation); unit: kJ/day
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
kJ/day | 1133.963 (1399.8793)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Test type: Superiority; p = 0.041, paired t-test

3. Secondary Outcome: Relative Change From Baseline in Actual Weekly Parenteral Support (PS) Volume at Weeks 4, 24, and 52
Description: The sum of daily PS volume (including extra fluids) from weekly PS diary data recorded for the corresponding analysis timepoint was used for analysis.
Time Frame: Baseline, Week 4, Week 24, and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change in PS volume
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
percentage change in PS volume
  Week 4 | -0.73 (2.709)
  Week 24 | -39.99 (22.588)
  Week 52 | -52.44 (29.192)

4. Secondary Outcome: Absolute Change From Baseline in Actual Weekly PS Volume at Weeks 24 and 52
Description: as for outcome 3
Time Frame: Baseline, Week 24 and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
mL
  Week 24 | -3510.000 (1893.7859)
  Week 52 | -4701.778 (2389.9652)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Week 24; Test type: Superiority; p < 0.001, paired t-test
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Week 52; Test type: Superiority; p < 0.001, paired t-test

5. Secondary Outcome: Number of Participants Who Achieved a Reduction of at Least 1 Day Per Week of PS From Baseline at Weeks 24 and 52
Description: Participants were considered to have a reduction of at least one day per week of PS from Baseline (incl. extra fluids) if the number of days with PS from weekly PS diary data recorded for the corresponding analysis timepoint was smaller compared to the number of days with PS from weekly PS diary data for Baseline.
Time Frame: Baseline, Week 24 and Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  Week 24 | 5
  Week 52 | 7

6. Secondary Outcome: Number of Participants Considered Clinical Responders at Weeks 24 and 52
Description: Clinical response was defined as a 20% reduction of PS volume from Baseline. The sum of daily PS volume (including extra fluids) from weekly PS diary data recorded for the corresponding analysis timepoint was used for analysis.
Time Frame: Baseline, Week 24 and 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  Week 24 | 7
  Week 52 | 9

7. Secondary Outcome: Number of Participants Who Achieved Enteral Autonomy at Weeks 24 and 52
Description: Enteral autonomy was defined as a participant not receiving PS for hydration or parenteral nutrition (PN) for calories. Participants may have still receive minimal fluid to maintain patency of the central line or for specific elemental/micro-nutrient needs (e.g., <100 mL fluid for administration of magnesium).
Time Frame: Weeks 24 and 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  Week 24 | 0
  Week 52 | 2

8. Secondary Outcome: Absolute Change in Total Energy in PN From Baseline at Weeks 24 and 52
Description: PN was defined as PS that includes protein, carbohydrate, fat, vitamins, and/or trace elements.
Time Frame: Baseline, Week 24 and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
kcal
  Week 24 | -2763.889 (1830.8065)
  Week 52 | -3510.111 (1927.2066)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Week 24; Test type: Superiority; p = 0.002, paired t-test
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Week 52; Test type: Superiority; p < 0.001, paired t-test

9. Secondary Outcome: Relative Change in Absorption of Energy Over MB Periods From Baseline at Week 48
Description: The absorption was defined as dietary intake minus output from fecal excretion over a 72-hour MB period at a given analysis time point. Since dietary intake and fecal excretion were measured daily, i.e., up to three measurements may contribute to absorption calculations, the average over all available daily absorption measurements over the 72-hour period were used for analysis.
Time Frame: Baseline and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
percentage change | 29.23 (36.898)

10. Secondary Outcome: Absolute Change in Absorption of Macronutrients Over MB Periods From Baseline at Weeks 4 and 48
Description: as for outcome 9
Time Frame: Baseline, Week 4 and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kJ/day
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
kJ/day
  Fat - Week 4 | 247.281 (661.1866)
  Fat - Week 48 | 406.741 (776.4802)
  Carbohydrate - Week 4 | 272.881 (675.1125)
  Carbohydrate - Week 48 | 877.011 (945.2279)
  Protein - Week 4 | 176.178 (280.0788)
  Protein - Week 48 | 194.400 (285.2597)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Fat absorption increase at Week 4; Test type: Superiority; p = 0.294, paired t-test
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Fat absorption increase at Week 48; Test type: Superiority; p = 0.155, paired t-test
Statistical Analysis 3: Comparison: Apraglutide SC Injections, Once Weekly; Carbohydrate absorption at Week 4; Test type: Superiority; p = 0.260, paired t-test
Statistical Analysis 4: Comparison: Apraglutide SC Injections, Once Weekly; Carbohydrate absorption at Week 48; Test type: Superiority; p = 0.024, paired t-test
Statistical Analysis 5: Comparison: Apraglutide SC Injections, Once Weekly; Protein absorption at Week 4; Test type: Superiority; p = 0.096, paired t-test
Statistical Analysis 6: Comparison: Apraglutide SC Injections, Once Weekly; Protein absorption at Week 48; Test type: Superiority; p = 0.075, paired t-test

11. Secondary Outcome: Absolute Change in Urine Volume Over MB Periods From Baseline at Week 4 and Week 48
Description: Based on average daily urine volume data derived as per balance period calculations.
Time Frame: Baseline, Week 4 and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
mL/day
  Week 4 | 246.889 (343.3609)
  Week 48 | -178.556 (299.5613)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Week 4; Test type: Superiority; p = 0.063, paired t-test
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Week 48; Test type: Superiority; p = 0.112, paired t-test

12. Secondary Outcome: Absolute Change in Absorption of Energy Over MB Periods From Baseline at Week 4
Description: as for outcome 9
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kJ/day
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
kJ/day | 494.259 (1355.5857)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Test type: Superiority; p = 0.306, paired t-test

13. Secondary Outcome: Absolute Change in Urinary Electrolytes Over MB Periods From Baseline at Week 4 and Week 48
Description: Since urinary electrolytes data were measured over the 72-hour MB period, the average of all available results were used for analyses for each MB parameter at a given analysis time point.
Time Frame: Baseline, Week 4 and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cmol/L
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
cmol/L
  Calcium - Week 4 | 0.1444 (1.09818)
  Calcium - Week 48 | -0.5532 (2.28264)
  Magnesium - Week 4 | -0.258 (0.8370)
  Magnesium - Week 48 | -2.306 (3.1400)
  Sodium - Week 4 | 31.668 (24.1946)
  Sodium - Week 48 | 17.097 (50.1676)
  Potassium - Week 4 | 2.047 (16.8154)
  Potassium - Week 48 | -8.012 (13.5798)
  Urea - Week 4 | 7.693 (59.2590)
  Urea - Week 48 | -89.649 (77.9786)
  Creatinine - Week 4 | 0.198 (1.0071)
  Creatinine - Week 48 | -0.011 (1.3283)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Calcium, Week 4; Test type: Superiority; p = 0.704, paired t-test; Median Difference (Final Values) = 0.3346, 95% CI 2-sided [-0.7887 to 0.8748] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Calcium, Week 48; Test type: Superiority; p = 0.488, paired t-test; Median Difference (Final Values) = -0.1040, 95% CI 2-sided [-2.7442 to 0.8896] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 3: Comparison: Apraglutide SC Injections, Once Weekly; Magnesium, Week 4; Test type: Superiority; p = 0.382, paired t-test; Median Difference (Final Values) = -0.219, 95% CI 2-sided [-0.896 to 0.313] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 4: Comparison: Apraglutide SC Injections, Once Weekly; Magnesium, Week 48; Test type: Superiority; p = 0.059, paired t-test; Median Difference (Final Values) = -1.566, 95% CI 2-sided [-5.279 to -0.165] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 5: Comparison: Apraglutide SC Injections, Once Weekly; Sodium, Week 4; Test type: Superiority; p = 0.004, paired t-test; Median Difference (Final Values) = 33.116, 95% CI 2-sided [5.510 to 51.861] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 6: Comparison: Apraglutide SC Injections, Once Weekly; Sodium, Week 48; Test type: Superiority; p = 0.337, paired t-test; Median Difference (Final Values) = 20.727, 95% CI 2-sided [-27.758 to 55.828] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 7: Comparison: Apraglutide SC Injections, Once Weekly; Potassium, Week 4; Test type: Superiority; p = 0.724, paired t-test; Median Difference (Final Values) = 1.618, 95% CI 2-sided [-11.870 to 14.931] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 8: Comparison: Apraglutide SC Injections, Once Weekly; Potassium, Week 48; Test type: Superiority; p = 0.115, paired t-test; Median Difference (Final Values) = -9.190, 95% CI 2-sided [-18.880 to 3.737] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 9: Comparison: Apraglutide SC Injections, Once Weekly; Urea, Week 4; Test type: Superiority; p = 0.707, paired t-test; Median Difference (Final Values) = 12.297, 95% CI 2-sided [-39.551 to 52.617] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 10: Comparison: Apraglutide SC Injections, Once Weekly; Urea, Week 48; Test type: Superiority; p = 0.009, paired t-test; Mean Difference (Final Values) = -91.487, 95% CI 2-sided [-159.956 to -20.068] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 11: Comparison: Apraglutide SC Injections, Once Weekly; Creatinine, Week 4; Test type: Superiority; p = 0.572, paired t-test; Median Difference (Final Values) = 0.281, 95% CI 2-sided [-0.649 to 0.960] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline
Statistical Analysis 12: Comparison: Apraglutide SC Injections, Once Weekly; Creatinine, Week 48; Test type: Superiority; p = 0.981, paired t-test; Median Difference (Final Values) = -0.136, 95% CI 2-sided [-1.060 to 1.073] — Based on one-sample (paired) Hodges-Lehmann median estimator for non-parametric estimate of change from baseline

14. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Inventory (PSQI) Total Score at Week 24 and Week 52
Description: The PSQI is a patient-reported questionnaire used to measure the quality and patterns of sleep, over the past month. The PSQI has seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. Minimum Score = 0 (better); Maximum Score = 21 (worse). A negative change from baseline represents an reduction in symptoms.
Time Frame: Baseline, Week 24 and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
score on a scale
  Week 24 | -1.89 (2.667)
  Week 52 | -1.56 (1.509)
Statistical Analysis 1: Comparison: Apraglutide SC Injections, Once Weekly; Week 24; Test type: Superiority; p = 0.066, paired t-test
Statistical Analysis 2: Comparison: Apraglutide SC Injections, Once Weekly; Week 52; Test type: Superiority; p = 0.015, paired t-test

15. Secondary Outcome: Change From Baseline in Patient Global Impression of Change (PGIC) at Week 24 and Week 52
Description: PGIC v2.0 is a single-item questionnaire using a 5-point verbal rating scale, to assess overall change in the participants status after taking the study drug. Response options range from 2= very much better to -2= very much worse.
Time Frame: Baseline, Week 24 and Week 52
Population: The full analysis set included all participants who received at least one dose of trial treatment and contributed at least one valid post-baseline efficacy point. Participants with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  Week 24: number analyzed (Participants) | 8
  Week 24: 2 (Much Better) | 6
  Week 24: 1 (A Little Better) | 2
  Week 52: 2 (Much Better) | 8
  Week 52: 1 (A Little Better) | 1

16. Secondary Outcome: Secondary: Patient Global Impression of Treatment Satisfaction (PGI-TS) at Week 24 and Week 52
Description: This form is a single-item questionnaire assessing the participant's satisfaction with the trial medication over the preceding 7 days. Response options range from -2 to 2, very dissatisfied to very satisfied.
Time Frame: Week 24 and Week 52
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
Participants
  Week 24: number analyzed (Participants) | 8
  Week 24: 2 (Very Satisfied) | 5
  Week 24: 1 (Satisfied) | 3
  Week 52: 2 (Very Satisfied) | 3
  Week 52: 1 (Satisfied) | 6

17. Secondary Outcome: Change From Baseline in Patient Global Impression of Satisfaction With Parenteral Support (PGI-SPS) at Week 24 and Week 52
Description: This is a single-item questionnaire assessing the participant's satisfaction with PS over the preceding 7 days. Response options range from -2 to 2, very dissatisfied to very satisfied. A reduction from baseline represents a decrease in satisfaction.
Time Frame: Baseline, Week 24 and Week 52
Population: The full analysis set included all participants who received at least one dose of trial treatment and contributed at least one valid post-baseline efficacy point. Partcipants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 5
score on a scale
  Week 24 | -0.20 (0.447)
  Week 52: number analyzed (Participants) | 4
  Week 52 | 0.00 (0.000)

18. Secondary Outcome: Change From Baseline in Patient Global Impression of Parenteral Support Impact (PGI-PSI) at Week 24 and Week 52
Description: This is a three-item questionnaire assessing the impact of PS on the participant's sleep, daily activities, and quality of life (QoL) over the past 7 days. All questions have response options ranging from 0 to 4, not at all to extremely. A reduction from baseline represents a decrease in symptoms.
Time Frame: Baseline, Week 24 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 5
score on a scale
  Sleep Impact: Week 24 | -0.40 (1.517)
  Sleep Impact: Week 52: number analyzed (Participants) | 4
  Sleep Impact: Week 52 | -0.50 (1.291)
  Daily Activities Impact: Week 24 | -0.80 (1.643)
  Daily Activities Impact: Week 52: number analyzed (Participants) | 4
  Daily Activities Impact: Week 52 | -1.00 (1.414)
  QoL Impact: Week 24 | -1.40 (1.140)
  QoL Impact: Week 52: number analyzed (Participants) | 4
  QoL Impact: Week 52 | -1.25 (0.957)

19. Secondary Outcome: Trough Apraglutide Plasma Concentration (Ctrough)
Time Frame: Pre-dose on Weeks 2, 4, 12, 24, 32, 40, 48, and 52
Population: The safety analysis set included all participants exposed to trial medication. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
ng/mL
  Week 2: number analyzed (Participants) | 4
  Week 2 | 1.928 (0.7058)
  Week 4: number analyzed (Participants) | 3
  Week 4 | 1.217 (0.2902)
  Week 12: number analyzed (Participants) | 5
  Week 12 | 1.934 (0.6665)
  Week 24: number analyzed (Participants) | 4
  Week 24 | 2.863 (1.0668)
  Week 32: number analyzed (Participants) | 7
  Week 32 | 1.739 (0.6805)
  Week 40: number analyzed (Participants) | 5
  Week 40 | 2.386 (0.9587)
  Week 48: number analyzed (Participants) | 3
  Week 48 | 3.810 (1.1031)
  Week 52 | 2.678 (1.4039)

20. Secondary Outcome: Mean Plasma Citrulline Level
Time Frame: Baseline and Weeks 2, 4, 12, 24, 32, 40, 48, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Apraglutide SC Injections, Once Weekly
Number analyzed (Participants) | 9
μmol/L
  Baseline | 11.571 (9.7091)
  Week 2 | 13.516 (9.8136)
  Week 4: number analyzed (Participants) | 8
  Week 4 | 15.531 (12.4055)
  Week 12 | 14.860 (12.2165)
  Week 24 | 14.810 (11.8877)
  Week 32 | 14.994 (12.6880)
  Week 40 | 17.860 (15.8020)
  Week 48 | 16.638 (14.9346)
  Week 52 | 14.714 (11.7896)

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 55 weeks
Description: The safety analysis set included all participants exposed to trial medication.
Arm/Group | Apraglutide SC Injections, Once Weekly
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apraglutide SC Injections, Once Weekly (N=9)
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Device dislocation (Product Issues) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apraglutide SC Injections, Once Weekly (N=9)
Haematoma (Vascular disorders) | 1
Asthenia (General disorders) | 1
Complication associated with device (General disorders) | 1
Catheter site irritation (General disorders) | 1
Injection site erythema (General disorders) | 2
Injection site pruritus (General disorders) | 1
Fatigue (General disorders) | 1
Injection site haematoma (General disorders) | 1
Injection site pain (General disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Weight decreased (Investigations) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Bone contusion (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Regurgitation (Gastrointestinal disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Influenza (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Vascular device infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 1
Asymptomatic COVID-19 (Infections and infestations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04964986/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04964986/SAP_001.pdf